CLINICAL TRIAL: NCT05664516
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Effects of Intranasal Oxytocin in Adults With Binge-eating Disorder
Brief Title: A Study of the Effects of Oxytocin in Adults With Binge-eating Disorder
Acronym: STROBE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Elizabeth Austen Lawson, Director, Interdisciplinary Oxytocin Research Program, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022P002727
Record Dates: First submitted 2022-12-16; First posted 2022-12-23 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-06

CONDITIONS: Binge-eating Disorder
Keywords: Binge; Binge-eating disorder; Oxytocin; Over-eating; Impulse Control
MeSH Terms: conditions — Binge-Eating Disorder; Hyperphagia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study staff and patients are blinded. The pharmacist is unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo Arm (Placebo Comparator): Solution without oxytocin
  Interventions: Drug: Placebo
- TNX-1900 (Experimental): Solution with oxytocin
  Interventions: Drug: TNX-1900 (Tonix Pharmaceuticals)

INTERVENTIONS:
Drug: TNX-1900 (Tonix Pharmaceuticals) — oxytocin nasal spray
  Arms: TNX-1900
Drug: Placebo — Nasal solution without oxytocin
  Arms: Placebo Arm

SUMMARY:
This study evaluates the impact of intranasal oxytocin vs placebo in patients with binge eating disorder or episodes of binging. We hypothesize that 8 weeks of intranasal oxytocin vs placebo will improve clinical outcomes [reduction in bingeing frequency], and have a satisfactory safety and tolerability profile. We will also explore the predictive value of changes in homeostatic appetite, reward sensitivity, and impulse control, the identified underlying mediators, as assessed 4 weeks into the intervention, for treatment success after 8 weeks of the intervention.

DETAILED DESCRIPTION:
Study staff will screen patients for eligibility as per eligibility criteria. At least 60 eligible patients will be randomized 1:1 (active oxytocin: placebo) by an unblinded pharmacist. All other study staff and test subjects will be blinded. Study subject medical histories, physical exams, anthropometric measurements, labs, EKG's, and eating habits will be monitored over 8 weeks. Subjects will be evaluated at the following intervals: Baseline, week 2, week 4, week 8, and week 16 (8 weeks post-treatment).

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18-70 years old
* BMI greater than or equal to 18.5
* BED as assessed by Structured Clinical Interview for DSM-5 Disorders (SCID-5-RV) OR Other Specified Feeding or Eating Disorder (OSFED) - Binge-eating disorder (of low frequency and/or limited duration) (SCID-5-RV) OR Bulimia Nervosa (BN) through excessive exercise and/or fasting to avoid gaining weight after episodes of binge eating. For individuals with OSFED-BED, the frequency of subjective and objective binge eating episodes will meet the frequency (Criterion D) for BED.

Exclusion Criteria:

* Substance use disorder active within the last 6 months, or clinical suspicion of ongoing substance use disorder at the discretion of the study clinician at the time of screening based on history and/or laboratory results
* Medication changes that have not reached steady state concentration, measured by the equivalent of 5 half-lives of that medication
* Use of medications for binge eating disorder or weight loss unless at a stable dose for at least 12 weeks
* History of any of the following medical conditions: inflammatory bowel disease; epilepsy; untreated thyroid disease
* History of known cardiovascular disease, including coronary artery disease, heart failure, reduced ejection fraction, hypertrophic cardiomyopathy, ventricular arrhythmias, or prolonged QT
* Hematocrit >2% below normal
* Hemoglobin A1c >8%
* Use of insulin
* ALT or AST >2.5 times upper limit of normal
* Glomerular filtration rate < 60 mL/min
* Hyponatremia. Note that, in order to be randomized, subjects must have Na ≥ 135 mEq/L.
* Pregnancy or breastfeeding
* Unwilling to use a medically acceptable form of contraception throughout the study period (female of child-bearing potential only)
* History of psychosis or active suicidal ideation
* Major depressive disorder likely to require initiation or change in active treatment
* Borderline personality disorder as assessed by the McLean Screening Instrument for Borderline Personality Disorder (MSI-BPD)
* Current nicotine use, unless stable use for at least 12 weeks.
* Participation in any clinical study involving an investigational drug, device, or biologic within 1 month of randomization
* Any significant illness, condition, or medication that the Investigator determines could interfere with study participation and impact data collection or subject safety

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Binge Frequency | 8 weeks
  Change in binge frequency as assessed by the Eating Disorder Examination clinical interview

SECONDARY OUTCOMES:
Reward sensitivity | 8 weeks
  Predictive value of 4-week change in reward sensitivity per the Temporal Experience of Pleasure Scale (TEPS) Anticipatory Experience of Pleasure subscale score for 8-week change in binge episodes. Higher scores=greater anticipatory pleasuure/less anhedonia. Minimum/Maximum: 10-60
Impulse control | 8 weeks
  Predictive value of 4 week change in impulse control per Stop-Signal Reaction time in a Stop-Signal Task for 8 week change in binge frequency

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Lawson, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Neuroendocrine Unit Research Center, Boston, Massachusetts, United States